CLINICAL TRIAL: NCT06656286
Title: Hysteroscopic Intrauterine Suturing by Using X-Tack - Pilot Study
Brief Title: Hysteroscopic Intrauterine Suturing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: EMC-0086-24
Record Dates: First submitted 2024-10-08; First posted 2024-10-24 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-10

CONDITIONS: Niche; Uterine Disease
MeSH Terms: conditions — Uterine Diseases | interventions — Hysteroscopes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Women undergoing laparoscopic hysterectomy (Experimental): Women undergoing laparoscopic hysterectomy for benign indication with no evidence or suspicious for malignancy.
  Interventions: Device: Intra-Uterine suturing by X-TACK device and hysteroscope

INTERVENTIONS:
Device: Intra-Uterine suturing by X-TACK device and hysteroscope — After general anesthesia and entering the abdomen with the laparoscope, Truclear hysteroscope with X-tack attached will be inserted to the uterine cavity. Insertion of normal saline to the cavity and applying 4 points suturing to the uterus. The procedure will be monitored by external laparoscopic camera located in the abdominal cavity. After the hysterectomy the uterus will be opened and the suture will be examine.
  A preoperative intrauterine incision using a hysteroscope, followed by suturing, will be considered based on the success of the first procedure.

SUMMARY:
Clinical trial The aim of the study is to evaluate the safety and feasibility of intrauterine suturing with Apollos X-tack, inserted into the uterus by hysteroscope.

Primary outcome:

Intrauterine suture will sustain the procedure - when the uterus will be opened the suture will be observed.

Secondary outcome:

Procedure complications. Study Design Interventional pilot Study

Study group:

Women undergoing laparoscopic hysterectomy.

DETAILED DESCRIPTION:
Introduction:

A hysteroscopy is a procedure used to examine and treat the inside of the uterus.

Apollo X-tack is an endoscopic apparatus for stomach defect closure by gastroscopy.

The aim of this study is to evaluate the safety and feasibility of intrauterine suturing with Apollos X-tack inserted into the uterus by hysteroscope.

Study Design Interventional pilot study

Study group:

Women undergoing laparoscopic hysterectomy.

Inclusion criteria:

Benign indication for hysterectomy

Exclusion from the study:

Evidence or suspicious for malignancy

Sample size calculation:

Pilot study of 2 patients.

Primary outcome:

Intrauterine suture will sustain the procedure - when the uterus will be opened the suture will be observed.

Secondary outcome:

Procedure complications.

Recruitment:

The recruitment of the patients will be done at the gynecology department before the surgery.

Procedure:

After general anesthesia and entering the abdomen with the laparoscope, Truclear hysteroscope with X-tack attached will be inserted to the uterine cavity. Insertion of normal saline to the cavity and applying 4 points suturing to the uterus. The procedure will be monitored by external laparoscopic camera located in the abdominal cavity. After the hysterectomy the uterus will be opened and the suture will be examine.

A preoperative intrauterine incision using a hysteroscope, followed by suturing, will be considered based on the success of the first procedure.

CRF:

Demographics information, obstetrics and gynecology information, surgery type, surgery indication.

Procedure duration, success, amount of fluid used, cervical dilatation, complications.

ELIGIBILITY:
Inclusion Criteria:

* Benign indication for hysterectomy

Exclusion Criteria:

* Evidence or suspicious for malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-04-25 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-07-02 (Estimated)

PRIMARY OUTCOMES:
Device Feasibility (intrauterine suturing) - The suture will sustain inside the uterus. | Immediately after the procedure.
  When the uterus will be opened the suture will be observed.

SECONDARY OUTCOMES:
Safety: Procedure complications - Uterine perforation, vaginal\cervical\uterine injury. | Immediately after the procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Emek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vila Famada A, Cos Plans R, Costa Canals L, Rojas Torrijos M, Rodriguez Vicente A, Bainac Albadalejo A. Outcomes of surgical hysteroscopy: 25 years of observational study. J Obstet Gynaecol. 2022 Jul;42(5):1365-1369. doi: 10.1080/01443615.2021.1971176. Epub 2021 Dec 16. PMID 34913810
- [Background] Umranikar S, Clark TJ, Saridogan E, Miligkos D, Arambage K, Torbe E, Campo R, Di Spiezio Sardo A, Tanos V, Grimbizis G; British Society for Gynaecological Endoscopy /European Society for Gynaecological Endoscopy Guideline Development Group for Management of Fluid Distension Media in Operative Hysteroscopy. BSGE/ESGE guideline on management of fluid distension media in operative hysteroscopy. Gynecol Surg. 2016;13(4):289-303. doi: 10.1007/s10397-016-0983-z. Epub 2016 Oct 6. No abstract available. PMID 28003797
- [Background] Bahar R, Shimonovitz M, Benshushan A, Shushan A. Case-control study of complications associated with bipolar and monopolar hysteroscopic operations. J Minim Invasive Gynecol. 2013 May-Jun;20(3):376-80. doi: 10.1016/j.jmig.2012.12.012. Epub 2013 Feb 27. PMID 23453765